CLINICAL TRIAL: NCT03089866
Title: Effect of Sedation on Cognitive Performance in the Elderly (Pilot Study)
Brief Title: Effect of Sedation on Cognitive Performance in the Elderly
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Froelich, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F141022006
Record Dates: First submitted 2017-03-07; First posted 2017-03-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Central nervous System; Memory functions; Executive functions; Cognitive impairment
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognitive Dysfunction | interventions — Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ASA Patients I or II: Participants are healthy (BMI <35), 55years and older, and have the ability to follow instructions. In this population we will quantify the effects of sedation with midazolam on auditory activation and cognitive performance (mini Mental State exam and complex reaction time).
  Interventions: Drug: Midazolam (0.02mg/kg)

INTERVENTIONS:
Drug: Midazolam (0.02mg/kg) — Quantify the effects of sedation with midazolam on auditory activation and cognitive performance (mini Mental State exam and complex reaction time).

SUMMARY:
The main goal of this study is to allow the anesthesiologist to make a more informed decision about the anesthetic requirement of a person prior to starting anesthesia. The preliminary data collected in this study will support a larger investigation aimed at gaining a better understanding of anesthetic susceptibility in general and in the elderly population which appears to be at greater risk for Postoperative Cognitive Dysfunction (POCD)

POCD is a short-term decline in cognitive function (especially in memory and executive functions) that may last from a few days to a few weeks after surgery. In rare cases, this disorder may persist for several months after major surgery. POCD is distinct from emergence delirium. It occurs most commonly in older patients and those with pre-existing cognitive impairment. POCD is common in adult patients of all ages at hospital discharge after major non-cardiac surgery, but only the elderly (aged 60 years or older) are at significant risk for long-term cognitive problems. The body's inflammatory response to surgery likely plays an important role, at least in elderly patients. Investigators also postulate that a relative 'anesthetic overdose' may be a significant risk factor. Hence, being able to make a better judgment on the dose needed for an individual is extremely important.

DETAILED DESCRIPTION:
Central nervous system (CNS) function is affected by sedation and anesthesia. This is evident from the desired clinical effects of sedative and anesthetic drugs. Recent evidence suggests that disruption CNS function may be prolonged and result in unwanted cognitive effects in predisposed individuals. Investigators know that there is a considerable pharmacokinetic (onset, distribution and elimination) and pharmacokinetic variability of neurotropic drugs even with in persons within a certain age and weight group. What the investigators do not know, is how to predict or quantify an individual's susceptibility to sedation and anesthesia and, more importantly, the potential cognitive susceptibility of an individual's brain to these drugs.

Auditory functional imaging is a well validated task. It can be applied as a short (5 minute) test. Investigators know (preliminary data) that the size of the brain activation area changes after sedation. Investigators now postulate that this change reflects a disruption of neuronal integration in the brain and that this change may be an objective measure of the cognitive effects of sedation for an individual.

As supportive data for an R-01 grant application the investigators propose to enroll 20 elderly subjects by public advertisement and quantify the effects of sedation with midazolam on auditory activation (auditory fMRI) and cognitive performance (mini Mental State exam and complex reaction time).

ELIGIBILITY:
Inclusion Criteria:

* Must be a healthy subject
* 55 years and older
* Able to follow study instructions.

Exclusion Criteria:

* Obesity (BMI > 35)
* Non-English speaking/reading
* Sleep apnea
* Moderate to severe bronchial asthma
* Cardiovascular problems including hypertension
* History of claustrophobia
* Presence of a pacemaker,
* Defibrillator,
* Any surgically placed metallic object,
* Presence of bullet or shrapnel in the body,
* Presence of a non-removable prosthetic,
* Use of a hearing aid if unable to hear otherwise,
* Head girth exceeding that of the head coil used in the MRI
* Extensive metal work on or in teeth
* Non-removable dentures or bridgework, epilepsy
* Chronic pain medication use/abuse
* Excessive tattoos (local skin heating can occur with tattoos containing ferromagnetic particles)
* History of surgery for which the details are unavailable
* Allergy to Midazolam
* History of drug abuse

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants classified by the American Society of Anesthesiologists (ASA) as a Class I or II patient.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Effect of a single dose of midazolam on cognitive function. | Baseline to 1hour
  Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores before and after sedation
Effect of a single dose of Midazolam on Auditory Activation | Baseline to 1 hour
  Change in Brain activation before and after sedation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Froelich, MD, Principal Investigator — Anesthesiology ad Perioperative Medicine
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bryson GL, Wyand A. Evidence-based clinical update: general anesthesia and the risk of delirium and postoperative cognitive dysfunction. Can J Anaesth. 2006 Jul;53(7):669-77. doi: 10.1007/BF03021625. PMID 16803914
- [Background] Folstein, Marshal F., Susan E. Folstein, and Paul R. McHugh.
- [Background] Wickelgren, Wayne A.
- [Background] Deary, Ian J., and Geoff Der.